CLINICAL TRIAL: NCT00050154
Title: An Open-Label, Phase 2 Study to Evaluate the Efficacy and Safety of the Farnesyl-Transferase Inhibitor ZARNESTRA(tm) (R115777) in Subjects With High-Risk Myelodysplastic Syndrome (MDS)
Brief Title: Study of Tipifarnib in Patients With High-Risk Myelodysplastic Syndrome (MDS)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR004027; NCT00722787 (obsolete NCT alias)
Record Dates: First submitted 2002-11-22; First posted 2002-11-25 (Estimated); Last update posted 2010-04-27 (Estimated); Status verified 2010-04

CONDITIONS: Myelodysplastic Syndrome
Keywords: R115777; Myelodysplastic syndromes; Tipifarnib; Zarnestra
MeSH Terms: conditions — Myelodysplastic Syndromes | interventions — tipifarnib

INTERVENTIONS:
Drug: ZARNESTRA, tipifarnib, R115777

SUMMARY:
The purpose of this study is to characterize the hematological response rate, as well as other parameters of efficacy and safety induced by tipifarnib in patients with high-risk myelodysplastic syndrome (MDS). Tipifarnib belongs to a class of drugs called Farnesyl Transferase Inhibitors (FTI). It blocks proteins that make cancer cells grow.

DETAILED DESCRIPTION:
Treatment with tipifarnib will be given during one or more periods of time called cycle(s). Each cycle will be 28 days long and patients will take tipifarnib for the first 21 days of each cycle. No medication will be taken during the last 7 days of each cycle. On day 1 and 15 of each cycle, patients will be asked about any side effects that have occurred since their last visit. Blood will drawn for routine testing to evaluate any possible effects of tipifarnib on white blood cells or on specific elements, that can be measured in the blood. The study doctor will decide if any bone marrow aspirates or biopsies should be taken. Tipifarnib will be given until the patient's disease worsens or they develop unacceptable side effects or until they withdraw consent to receive tipifarnib. When tipifarnib treatment is ended or if the patient leaves the study early, they will be asked to come in for a final visit. The study doctor will decide if any blood draws, bone marrow aspirates or biopsies need to be taken.

Tipifarnib is 300 mg administered orally as three 100 mg tablets twice daily for the first 21 days in each 28-day cycle. Tipifarnib will be administered until the patient discontinues treatment due to disease progression or unacceptable toxicity.

ELIGIBILITY:
Inclusion Criteria:

* Pathological evidence of MDS
* Not more than 1 prior cytotoxic treatment for MDS
* Able to take oral study drug
* Able to understand and provide signed informed consent

Exclusion Criteria:

* Refractory anemia (RA) or RA with excess of blasts (RAEB) or patients with RAEB with < or = 10% marrow blasts
* Treatment-related MDS, if treated with chemotherapy less than 3 years ago
* Not adequately recovered from any treatment-related non-hematological toxicity
* Refractory to platelet transfusion
* Candidates for hematopoietic stem cell transplantation
* Previous therapy with a farnesyl transferase inhibitor
* Prior extensive radiation therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2002-07; Study Completion 2006-05 (Actual)

PRIMARY OUTCOMES:
The purpose of this research study is to determine if tipifarnib leads to a complete response for in patients with high-risk Myelodysplastic Syndrome (MDS).

SECONDARY OUTCOMES:
Efficacy will be assessed by evaluation of bone marrow and hematologic laboratory tests. Safety will be assessed by evaluation of adverse events and clinical laboratory tests.

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research and Development, L.L.C. Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.